CLINICAL TRIAL: NCT00793429
Title: A Double-Blind, Placebo-Controlled, Two-Way Cross-Over in Healthy Volunteers, to Evaluate the Pharmacokinetics, Tolerability and Cardiac Safety of Prucalopride at Steady-State
Brief Title: Safety Study of Prucalopride in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Movetis (Industry)
Other Study IDs: GBR-9
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2008-11-21 (Estimated); Status verified 2008-11

CONDITIONS: Healthy
Keywords: electrocardiographic safety; pharmacokinetics
MeSH Terms: interventions — prucalopride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Prucalopride
Other: Placebo

SUMMARY:
In this study healthy volunteers received increasing doses of prucalopride to study the tolerability and cardiac safety of prucalopride. The study hypothesis was that prucalopride at doses up to 10 mg has no clinically relevant effect on the cardiovascular safety in healthy volunteers.

DETAILED DESCRIPTION:
Single-centre, double-blind, placebo-controlled, cross-over study in 33 healthy volunteers with 2 sessions. Each session consisted of a run-in day for baseline assessments, 8 treatment days and 5 additional days for followup assessments. Subjects were randomised to start with either the prucalopride or placebo session. The prucalopride dose was consecutively escalated in 2 mg steps per day, starting from 2 mg up to 10 mg once daily If a subject did not tolerate the 10- or 8-mg dose, 1 step back in the dosage scheme was allowed, from 10 to 8 mg on Day 6, or from 8 to 6 mg on Day 5. Subjects with intolerance for doses of less than 6 mg, were withdrawn from the study. Repeated dosing (6, 8 or 10 mg) was continued once daily until Day 8, to achieve steady-state. During placebo, the number of placebo tablets was consecutively escalated in an identical way as described for prucalopride. Between the 2 sessions, there was a washout period of 14 to 21 days, to avoid any carry-over effect.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 45 years.
* Normal weight.
* Healthy on the basis of a pre-study physical examination, medical history, anamnesis,ECG, 24-hour Holter monitoring, echocardiogram and the results of blood biochemistry and haematology tests and a urinalysis carried out in 3 weeks preceding randomisation.

Exclusion Criteria:

* History or suspicion of alcohol, barbiturate, amphetamine or narcotic abuse.
* Smoking more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 6 months prior to selection.
* History of cardiac arrhythmias, bronchospastic or cardiovascular disease (e.g. ischaemic heart disease or cerebrovascular accident), diabetes mellitus, thyrotoxicosis,Parkinsonism.
* Presence of prolonged QTc (Bazett) on ECG at screening (QTc >450 ms in male subjects, QTc >470 ms in female subjects).
* Use of concomitant medication, except for oral contraceptives and paracetamol.
* Participation in an investigational drug study in 30 days prior to the first visit.
* Donation of blood in the 60 days preceding the first visit.
* Pregnancy or breast-feeding female.
* Female subjects of childbearing potential without adequate contraceptive protection during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult